CLINICAL TRIAL: NCT00486161
Title: Evaluation of Acylated Ghrelin Response Following Acute Exercise in Relation to Adiposity, Metabolic Homeostasis and Growth Hormone Secretion
Brief Title: Acylated Ghrelin Response to Acute Exercise in Obesity
Acronym: aeroghre
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Other Study IDs: 18C403
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Obesity
Keywords: Obesity; Ghrelin; Non-esterified fatty acids; Growth hormone; Insulin; Cycloergometer exercise
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Ghrelin is a GH-secretagogue gastrointestinal hormone that regulates feeding behavior by interacting directly with hypothalamic centers in concert with other negative and permissive neuromodulators. Ghrelin is involved in controlling energy balance in the short-term and long-term, and its levels are inversely related to the degree of obesity, insulin-resistance and energy accumulation. Consequently, obesity bears decreased ghrelin levels which increase upon weight loss, energy depletion and long-term exercise programs. Nevertheless, the role of acute exercise on the secretion of the bioactive component of ghrelin is yet unknown in conditions of normal and excessive body weight.

Our study examines acylated and total ghrelin secretion following a cycloergometric exercise test in obese and age- and sex-matched lean subjects to document if ghrelin components change as a function of fat accumulation, insulin homeostasis, growth hormone secretion, non-esterified fatty acid availability and exercise performance. Our study aims at testing the hypothesis that ghrelin components may be regulated by acute exercise, with concentrations at the exercise peak being related to acute metabolic homeostasis. Targetting this purpose may help to clarify ghrelin involvement in acute conditions unrelated to gastrointestinal activities.

DETAILED DESCRIPTION:
1. Ghrelin is the natural ligand of the hypothalamic GH-secretagogue receptor (GHS-R)-1a (1). Over the time, it has been documented that ghrelin predominantly functions as a central modulator of energy homeostasis via NP-Y and AgRP-containing neurons located in the arcuate nucleus of the hypothalamus (2). It thus promotes the drive to eat and governs long-term energy accumulation; clearly, circulating ghrelin concentrations are related to energy balance based on the following evidences (3):

   * ghrelin levels are acutely modulated by food intake and glucose administration
   * long-term ghrelin homeostasis reflects adiposity, insulin resistance and chronic exercise
   * in fasting and postabsorptive conditions, a negative correlation exists between ghrelin and resting energy expenditure independent of variations in insulin levels, energy intake, body composition or body weight.

   In summary, circulating ghrelin levels are approximately 30% lower than normal; are inversely related to increasing body fat, leptin and insulin levels; and are far less responsive to post-meal inhibition than in controls (3).
2. In the circulation, ghrelin is found as acylated and desacylated peptide. Ser(3)-octanoylation is a prerequisite for ghrelin biological activity (3). Des-octanoyl ghrelin variants have been additionally identified (4,5) and found to exert novel antiapoptotic effects in primary adult and cultured rat cardiomyocytes (6). Using specific immunoassays recognizing active (N-terminus) and total (N- plus C-terminus) ghrelin levels, assessment of circulating ghrelin concentrations helped to further discriminate specific functions of each at the hypothalamic level (7), on insulin sensitivity (8) or after bariatric surgery (9). Also, an association has been documented between obesity and total and acylated ghrelin concentrations, being respectively 30% and 56% lower than normal (10). Our laboratory showed previously that stratification of obese patients by the ratio of measured/predicted resting energy expenditure, allowed to detect a positive relationship between acylated ghrelin levels and the efficiency of energy expenditure (10). Speculatively, this could be interpreted as an obesity-related compensatory mechanism acting to contain the orexigenic signals afferent to the brain.
3. Studies on ghrelin responsiveness to cycloergometer exercise, treadmill exercise or long-distance marathons, originally showed no variation of ghrelin secretion (11-13). More recently, significant decrements of ghrelin levels following acute exercise bouts has been observed in elite athletes and their healthy controls, as well as in lean individuals (14, 15). While these findings suggested a link of ghrelin suppression with GH rise on one side and appetite regulation upon exercise on the other, little is known on the metabolic mechanisms regulating ghrelin response to acute exercise in the lean and obese state.

Based on these observations, our comparative study aims at exploring the response of ghrelin components to a standardized maximal exercise test in the lean and obese state, to identify the neuroendocrine and metabolic predictors of ghrelin response in these groups and document if ghrelin components change as a function of fat accumulation, insulin homeostasis, growth hormone secretion, non-esterified fatty acid availability and exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* healthy status
* lean (BMI < 25 kg/m2) and obese subjects (BMI>30 kg/m2)

Exclusion Criteria:

* cardiovascular disease
* gastrointestinal disease
* diabetes mellitus
* alcohol consumption (wine or equivalents) > 125 ml Day
* physical inability

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2004-03; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Marzullo, MD, PhD, Principal Investigator — Division of General Medicine
Locations (1):
- IRCCS Istituto Auxologico Italiano, Ospedale San Giuseppe, Piancavallo Di Oggebbio, Verbania, Italy

REFERENCES:
- [Background] Kojima M, Hosoda H, Date Y, Nakazato M, Matsuo H, Kangawa K. Ghrelin is a growth-hormone-releasing acylated peptide from stomach. Nature. 1999 Dec 9;402(6762):656-60. doi: 10.1038/45230. PMID 10604470
- [Background] Shintani M, Ogawa Y, Ebihara K, Aizawa-Abe M, Miyanaga F, Takaya K, Hayashi T, Inoue G, Hosoda K, Kojima M, Kangawa K, Nakao K. Ghrelin, an endogenous growth hormone secretagogue, is a novel orexigenic peptide that antagonizes leptin action through the activation of hypothalamic neuropeptide Y/Y1 receptor pathway. Diabetes. 2001 Feb;50(2):227-32. doi: 10.2337/diabetes.50.2.227. PMID 11272130
- [Background] van der Lely AJ, Tschop M, Heiman ML, Ghigo E. Biological, physiological, pathophysiological, and pharmacological aspects of ghrelin. Endocr Rev. 2004 Jun;25(3):426-57. doi: 10.1210/er.2002-0029. PMID 15180951
- [Background] Ariyasu H, Takaya K, Hosoda H, Iwakura H, Ebihara K, Mori K, Ogawa Y, Hosoda K, Akamizu T, Kojima M, Kangawa K, Nakao K. Delayed short-term secretory regulation of ghrelin in obese animals: evidenced by a specific RIA for the active form of ghrelin. Endocrinology. 2002 Sep;143(9):3341-50. doi: 10.1210/en.2002-220225. PMID 12193546
- [Background] Baldanzi G, Filigheddu N, Cutrupi S, Catapano F, Bonissoni S, Fubini A, Malan D, Baj G, Granata R, Broglio F, Papotti M, Surico N, Bussolino F, Isgaard J, Deghenghi R, Sinigaglia F, Prat M, Muccioli G, Ghigo E, Graziani A. Ghrelin and des-acyl ghrelin inhibit cell death in cardiomyocytes and endothelial cells through ERK1/2 and PI 3-kinase/AKT. J Cell Biol. 2002 Dec 23;159(6):1029-37. doi: 10.1083/jcb.200207165. Epub 2002 Dec 16. PMID 12486113
- [Background] Ghigo E, Broglio F, Arvat E, Maccario M, Papotti M, Muccioli G. Ghrelin: more than a natural GH secretagogue and/or an orexigenic factor. Clin Endocrinol (Oxf). 2005 Jan;62(1):1-17. doi: 10.1111/j.1365-2265.2004.02160.x. PMID 15638864
- [Background] St-Pierre DH, Karelis AD, Coderre L, Malita F, Fontaine J, Mignault D, Brochu M, Bastard JP, Cianflone K, Doucet E, Imbeault P, Rabasa-Lhoret R. Association of acylated and nonacylated ghrelin with insulin sensitivity in overweight and obese postmenopausal women. J Clin Endocrinol Metab. 2007 Jan;92(1):264-9. doi: 10.1210/jc.2006-1603. Epub 2006 Oct 24. PMID 17062757
- [Background] Korner J, Bessler M, Cirilo LJ, Conwell IM, Daud A, Restuccia NL, Wardlaw SL. Effects of Roux-en-Y gastric bypass surgery on fasting and postprandial concentrations of plasma ghrelin, peptide YY, and insulin. J Clin Endocrinol Metab. 2005 Jan;90(1):359-65. doi: 10.1210/jc.2004-1076. Epub 2004 Oct 13. PMID 15483088
- [Background] Marzullo P, Verti B, Savia G, Walker GE, Guzzaloni G, Tagliaferri M, Di Blasio A, Liuzzi A. The relationship between active ghrelin levels and human obesity involves alterations in resting energy expenditure. J Clin Endocrinol Metab. 2004 Feb;89(2):936-9. doi: 10.1210/jc.2003-031328. PMID 14764817
- [Background] Dall R, Kanaley J, Hansen TK, Moller N, Christiansen JS, Hosoda H, Kangawa K, Jorgensen JO. Plasma ghrelin levels during exercise in healthy subjects and in growth hormone-deficient patients. Eur J Endocrinol. 2002 Jul;147(1):65-70. doi: 10.1530/eje.0.1470065. PMID 12088921
- [Background] Schmidt A, Maier C, Schaller G, Nowotny P, Bayerle-Eder M, Buranyi B, Luger A, Wolzt M. Acute exercise has no effect on ghrelin plasma concentrations. Horm Metab Res. 2004 Mar;36(3):174-7. doi: 10.1055/s-2004-814342. PMID 15057671
- [Background] Kraemer RR, Durand RJ, Acevedo EO, Johnson LG, Kraemer GR, Hebert EP, Castracane VD. Rigorous running increases growth hormone and insulin-like growth factor-I without altering ghrelin. Exp Biol Med (Maywood). 2004 Mar;229(3):240-6. doi: 10.1177/153537020422900304. PMID 14988516
- [Background] Vestergaard ET, Dall R, Lange KH, Kjaer M, Christiansen JS, Jorgensen JO. The ghrelin response to exercise before and after growth hormone administration. J Clin Endocrinol Metab. 2007 Jan;92(1):297-303. doi: 10.1210/jc.2006-1435. Epub 2006 Oct 10. PMID 17032714
- [Background] Broom DR, Stensel DJ, Bishop NC, Burns SF, Miyashita M. Exercise-induced suppression of acylated ghrelin in humans. J Appl Physiol (1985). 2007 Jun;102(6):2165-71. doi: 10.1152/japplphysiol.00759.2006. Epub 2007 Mar 8. PMID 17347386
- [Derived] Marzullo P, Salvadori A, Brunani A, Verti B, Walker GE, Fanari P, Tovaglieri I, De Medici C, Savia G, Liuzzi A. Acylated ghrelin decreases during acute exercise in the lean and obese state. Clin Endocrinol (Oxf). 2008 Dec;69(6):970-1. doi: 10.1111/j.1365-2265.2008.03275.x. Epub 2008 Apr 14. No abstract available. PMID 18419786
- See also: Institution's description of scientific activities — http://www.auxologico.it